CLINICAL TRIAL: NCT04119505
Title: Pronostic Value of Diaphragmatic Excursion Measurement in Patients With Acute Respiratory Failure in the ED.
Brief Title: Value of Diaphragmatic Motion Measurement at Ultrasonography to Predict Poor Prognosis in Emergency Department Patients With Acute Respiratory Failure
Acronym: PREDIRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Poitiers University Hospital (Other); University Hospital, Brest (Other); Nord-Vienne Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0141
Record Dates: First submitted 2019-09-25; First posted 2019-10-08 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Dyspnea; Acute Respiratory Failure
Keywords: Diaphragmatic Excursion; Diaphragmatic Dysfunction; Emergency Department; Respiratory insufficiency; Acute respiratory failure
MeSH Terms: conditions — Dyspnea; Emergencies; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory failure is one of the most common diagnosis in patients admitted in the Emergency Department. Acute respiratory failure is associated with morbidity and mortality. Fifteen percent of patient will require ventilatory support and among them 40% will die.

Measurement of diaphragmatic motion (excursion) at ultrasonography is a noninvasive measure, allowing to assess diaphragm dysfunction. It could be useful in predicting poor prognosis in ED patients with respiratory failure .

In this study the investigators will compare the prognostic value of diaphragmatic excursion measurement at ultrasonography to that of the National Early Warning Score (NEWS) 2 in patients presenting with acute respiratory failure in the ED

The Investigators made the hypothesis that measurement of diaphragmatic excursion in ED patients with acute respiratory failure could be of value in predicting the need for ventilatory support or mortality within 28 days from ED admission

DETAILED DESCRIPTION:
Diaphragmatic dysfunction can be explored by measuring diaphragmatic excursion using ultrasonography in spontaneous ventilation patients.

Patients in spontaneous ventilation will undergo both diaphragmatic excursion measurement at ultrasonography and assessment of the News2 score as part of standard care.

ELIGIBILITY:
Inclusion criteria:

* Age equal or over 18 y.o
* Signs of acute respiratory failure defined by RR equal or over 25 br/min and/or signs of increased work of breathing
* Patients on spontaneous breathing

Exclusion criteria:

* Medical history of diaphragmatic dysfunction including stroke or diaphragmatic paralysis
* Patients on ventilatory support at ED admission or prior to inclusion
* Patients treated with curare
* Trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in the Emergency Department for Acute Respiratory Failure
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 28 days
  Adverse events are defined as a composite of mortality and/or cardiac arrest and/or need for ventilatory support (including invasive and/or noninvasive ventilation and/or high flow nasal cannula therapy) within 28 days from ED admission.

SECONDARY OUTCOMES:
Delay to initiation of ventilatory support | at day 28
  Ventilatory support is defined as invasive mechanical ventilation or non invasive ventilation or high-flow nasal cannula
Number of patients with adverse events at ED discharge | through ED stay (up to a day)
  Adverse events are defined as a composite of mortality and/or cardiac arrest and/or need for ventilatory support (including invasive and/or noninvasive ventilation and/or high flow nasal cannula therapy).
Number of patients with adverse events at hospital discharge | through hospital stay (up to a week)
  Adverse events are defined as a composite of mortality and/or cardiac arrest and/or need for ventilatory support (including invasive and/or noninvasive ventilation and/or high flow nasal cannula therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MARJANOVIC, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC